CLINICAL TRIAL: NCT00118482
Title: A Randomized Clinical Trial of Fludrocortisone for Vasovagal Syncope: The Second Prevention of Syncope Trial (POST II)
Brief Title: Clinical Trial for the Prevention of Vasovagal Syncope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Bob Sheldon, Professor of Cardiac Sciences, Medicine and Medical Genetics, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 130312; ISRCTN51802652
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Syncope, Vasovagal, Neurally-Mediated
Keywords: vasovagal syncope; randomized clinical trial; quality of life
MeSH Terms: conditions — Syncope, Vasovagal | interventions — fludrocortisone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fludrocortisone acetate (Experimental)
  Interventions: Drug: fludrocortisone acetate
- Placebo (Placebo Comparator)
  Interventions: Drug: fludrocortisone acetate

INTERVENTIONS:
Drug: fludrocortisone acetate — Fludrocortisone acetate to a maximum of 0.2 mg daily Placebo to a maximum of 0.2 mg daily

SUMMARY:
The main question in the study is whether people taking fludrocortisone are less likely to faint than people taking an inactive pill called a placebo.

Fludrocortisone is a drug that stimulates the body to retain salt and water. The investigators know from some studies that it might prevent people from fainting at home and in the community, while they are carrying on with their lives. There is some evidence that salt and water retention help prevent fainting, but no one has a clear idea about whether this is true. This study will try to determine if that is true.

DETAILED DESCRIPTION:
About 10% of adults faint recurrently. These patients are often highly symptomatic, have problems with employment and driving, and have well-documented reduced quality of life. There are no therapies that have withstood the test of adequately conducted and credible randomized clinical trials.

There is ample evidence of the importance of blood volume in the pathophysiology of vasovagal syncope. Fludrocortisone acetate is a corticosteroid with a mild enhancement of glucocorticoid activity and a marked increase in mineralocorticoid activity. It has no appreciable glucocorticoid effect at doses between 0.05 to 0.2 mg, which are the commonly used clinical doses for various disorders requiring mineralocorticoid adrenal replacement. The acute actions of fludrocortisone acetate are sodium and water retention, at the expense of urinary potassium excretion. Blood volume expansion with either dietary salt supplementation or fludrocortisone is often recommended by clinicians for the treatment of vasovagal syncope despite a paucity of good evidence for their efficacy. Four clinical studies suggest its utility in the prevention of syncope. Fludrocortisone might decrease the incidence of vasovagal syncope, but the quality of the evidence supporting its use is poor. There are no randomized, placebo-controlled trials of fludrocortisone for the prevention of vasovagal syncope. In this 5-year study the investigators will test the hypothesis that fludrocortisone prevents recurrences of vasovagal syncope.

ELIGIBILITY:
Inclusion Criteria:

* Syncope as a cause of loss of consciousness according to European Society of Cardiology criteria
* > 2 lifetime syncopal spells preceding enrollment
* > or = to -2 points on the Syncope Symptom Score for Structurally Normal Hearts
* Age > 18 years with informed consent, or age > 14 years with consent and informed parental consent

Exclusion Criteria:

* Other causes of syncope, such as ventricular tachycardia, complete heart block, postural (orthostatic) hypotension or hypersensitive carotid sinus syndrome
* An inability to give informed consent
* Important valvular, coronary, myocardial or conduction abnormality or significant arrhythmia
* Hypertrophic cardiomyopathy
* A known intolerance to fludrocortisone
* Another clinical need for fludrocortisone that cannot be met with other drugs
* A permanent pacemaker
* A seizure disorder
* A major chronic non cardiovascular disease
* Hypertension (blood pressure ≥ 130/85 on 2 occasions) or heart failure
* Renal dysfunction (baseline glomerular filtration rate reduced below 60 ml/min/1.73m2 according to the Cockroft-Gault formula)
* Diabetes mellitus
* Hepatic disease
* Glaucoma
* Any prior use of fludrocortisone acetate
* A 5-minute stand test resulting in diagnosis of postural orthostatic tachycardia syndrome or orthostatic hypotension

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2005-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Sheldon, MD PhD, Principal Investigator — University of Calgary, Faculty of Medicine
Locations (14):
- United States (3):
  - Boston University, Boston, Massachusetts
  - Vanderbilt University, Nashville, Tennessee
  - Virginia Cardiovascular Specialists, Richmond, Virginia
- Canada (11):
  - University of Calgary, Faculty of Medicine, Calgary, Alberta
  - Alberta Children's Hospital, Calgary, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II, Halifax Infirmary, Halifax, Nova Scotia
  - McMaster University, Hamilton Health Sciences, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University of Western Ontario, London Health Sciences, London, Ontario
  - University of Ottawa, Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Hopital Sacre Coeur de Montreal, Montreal, Quebec

REFERENCES:
- [Derived] Tan VH, Ritchie D, Maxey C, Sheldon R; POST Investigators. Prospective Assessment of the Risk of Vasovagal Syncope During Driving. JACC Clin Electrophysiol. 2016 Apr;2(2):203-208. doi: 10.1016/j.jacep.2015.10.006. Epub 2015 Nov 17. PMID 29766871
- [Derived] Sheldon R, Raj SR, Rose MS, Morillo CA, Krahn AD, Medina E, Talajic M, Kus T, Seifer CM, Lelonek M, Klingenheben T, Parkash R, Ritchie D, McRae M; POST 2 Investigators. Fludrocortisone for the Prevention of Vasovagal Syncope: A Randomized, Placebo-Controlled Trial. J Am Coll Cardiol. 2016 Jul 5;68(1):1-9. doi: 10.1016/j.jacc.2016.04.030. PMID 27364043
- [Derived] Raj SR, Rose S, Ritchie D, Sheldon RS; POST II Investigators. The Second Prevention of Syncope Trial (POST II)--a randomized clinical trial of fludrocortisone for the prevention of neurally mediated syncope: rationale and study design. Am Heart J. 2006 Jun;151(6):1186.e11-7. doi: 10.1016/j.ahj.2006.03.013. PMID 16781217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between October 1998 and April 2003 from university hospitals in Canada, Columbia, the United States and Poland.
Period: Overall Study
Arm/Group | Fludrocortisone Acetate | Placebo
Started | 105 (3 patients signed the consent but did not take the study medication.) | 105
Completed | 75 (210 in the Intention To Treat analysis) | 76
Not Completed | 30 | 29
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 23 | 22

BASELINE CHARACTERISTICS:
Population: Median age was 30.5 years and 146 were women.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fludrocortisone Acetate | Placebo | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Continuous [Median (Standard Deviation); unit: years] | 28 (11.5) | 31 (12) | 30.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 75 | 146
  Male | 34 | 30 | 64
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
  Canada | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be the Recurrence of Syncope in Follow up Period.
Description: This will be measured in terms of number of patients that had at least 1 syncopal spell in the 12 month follow up period.
Time Frame: Within 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fludrocortisone Acetate | Placebo
Number analyzed (Participants) | 105 | 105
Participants | 42 | 54

2. Secondary Outcome: The Frequency of Syncope Will be the First Secondary Outcome Measure.
Description: Frequency will be reported as 12- month syncope event rates (%)
Time Frame: Within 12 months
Measure: Mean (95% Confidence Interval); unit: rate %
Arm/Group | Fludrocortisone Acetate | Placebo
Number analyzed (Participants) | 105 | 105
rate % | 44.0 [42 to 94] | 60.5 [46 to 103]

3. Secondary Outcome: Presyncope Frequency, Duration, and Intensity Will be the Second Secondary Outcome Measures, Both Alone and in a Composite Score.
Time Frame: Within 12 months
Population: Data not analyzed because of variability of data collected on presyncope
Arm/Group | Fludrocortisone Acetate | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Quality of Life Will be the Third Secondary Outcome Measure. The Investigators Will Compare the Quality of Life in Treated and Untreated Patients.
Description: Quality of life will be the third secondary outcome measure. The investigators will compare the quality of life in patients on fludrocortisone vs placebo. Reported as RAND36 (Research ANd Development) score. The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Min value = 0 , Maximum value = 100. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fludrocortisone Acetate | Placebo
Number analyzed (Participants) | 76 | 85
score on a scale | 69 (21) | 84 (11)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the length of each participant's time in the trial up to 1 year.
Arm/Group | Fludrocortisone Acetate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 8/105 | 8/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludrocortisone Acetate (N=105) | Placebo (N=105)
Headache (General disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No